CLINICAL TRIAL: NCT04907448
Title: Optimization of Weight-bearing- and Walking-symmetry and Dynamic Balance Using an Isokinetic Strength Training Protocol in Children With Hemiparetic Cerebral Palsy
Brief Title: Isokinetic Strength Training in Children With Hemiparetic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0018/0062
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: A prospective pre-test post-test randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blind to the allocation of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IsoK-ST group (Experimental): Participants in this group received the usual physical rehabilitation program in addition to an IsoK-ST program.
  Interventions: Other: Physical Therapy
- Control group (Active Comparator): Participants in this group received the usual physical rehabilitation program only.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — The IsoK-ST group received their usual physical therapy program for 45 minutes, three times a week for eight successive weeks, which comprised advanced balance training, weight-bearing exercises, gait training, postural and flexibility exercises, and strength training exercises.
  Additionally, the IsoK-ST group received an IsoK-ST program, thrice/week for eight successive weeks.
  The control group received the usual physical rehabilitation program only for 45 minutes, three times a week for eight successive weeks.

SUMMARY:
This study endeavored to assess the effect of an isokinetic strength training (IsoK-ST) program on weight-bearing symmetry, gait-symmetry, and dynamic balance in children with hemiparetic cerebral palsy (HCP). Thirty-six children with HCP were randomly allocated to the IsoK-ST group (n = 18, received their usual physical rehabilitation program plus an IsoK-ST program) or the Control group (n =18, received usual physical rehabilitation alone). Both groups were assessed for weight-bearing symmetry, gait-symmetry, and dynamic balance before and after treatment.

DETAILED DESCRIPTION:
Thirty-six children with HCP were recruited from the Physical Therapy Outpatient Clinic of Collee of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, King Khalid Hospital, and a tertiary referral hospital, Al-Kharj, Saudi Arabia. Their age ranged between 8 and 16 years, were functioning at levels I or II according to the Gross Motor Function Classification System, and had spasticity level 1 or 1+ per the Modified Ashworth Scale. Children were excluded if they had structural nonreducible deformities, underwent neuromuscular or orthopedic surgery in the last 12 months, submitted to BOTOX injection in the past 6 months, sensory-perceptual disorders, unstable convulsions, cardiopulmonary problems preventing them from performing high-intense exercise training.

Outcome measures

1. Weight-bearing symmetry index: The weight-bearing symmetry index for the rearfoot and forefoot segments were assessed through a pressure analysis system
2. Gait-symmetry Indices: Gait symmetry indices (Spatial and temporal) were measured through the portable GAIT Rite system.
3. Dynamic balance: The directional dynamic limit of stability (forward, backward, paretic, and non-paretic) and overall limit of stability were assessed using the Biodex balance system.

The IsoK-ST and control groups received their usual physical rehabilitation program for 45 minutes, three times a week for eight consecutive weeks. The program comprised advanced balance training, and gait training exercises, postural and flexibility exercises, strength training exercises. Additionally, the IsoK-ST group received an IsoK-ST program, thrice/week for eight weeks per the National Strength and Conditioning Association guidelines and American Academy of Pediatrics safety standards. The IsoK-ST consisted of 3 sets (5-10 repetitions) of maximal concentric contraction of knee extensors and flexors on the affected side at angular speeds of 90, 120, 180, and 240 deg./sec., with intervals of rest for two minutes after each selected speed. The IsoK-ST workout was proceeded by a 5-minute warm-up and ended up with a 5-minute cool-dowm.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparetic cerebral palsy
* Age 8-16 years
* Motor function level I or II according to the Gross Motor Function Classification System.
* Spasticity level 1 or 1+ according to the Modified Ashworth Scale

Exclusion Criteria:

* Structural deformities
* Musculoskeletal or neural surgery in the last year
* BOTOX injection in the last 6 months.
* Cardiopulmonary disorders interfering with the ability to engage in exercise training.
* Hemispatial neglect.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2018-12-23 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Weight-bearing symmetry | 2 months
  The weight-bearing symmetry indices of the rearfoot and forefoot segments were measured using a Pressure analysis system.
Gait-symmetry indices | 2 months
  Gait symmetry indices (spatial and temporal) were measured about the step length and single-limb support time of the paretic and non-paretic leg through the portable GAIT Rite system
Dynamic balance | 2 months
  The directional (forward, backward, paretic, and non-paretic) and overall dynamic limits of stability were assessed through the Biodex balance system.

CONTACTS AND LOCATIONS:
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No